CLINICAL TRIAL: NCT03057483
Title: Active Surveillance for Adverse Events Following Immunization With the Trivalent Influenza Vaccine (Split Virion and Inactivated) Produced at Butantan Institute
Brief Title: Active Surveillance for Adverse Events Following Immunization With the Influenza Vaccine Produced at Butantan Institute
Acronym: FLU-05-IB
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: FLU-05-IB
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-07

CONDITIONS: Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Elderly: People over 60 years of age. seasonal influenza vaccine
  Interventions: Biological: Seasonal Influenza vaccine
- Health care workers: People working in health care services seasonal influenza vaccine
  Interventions: Biological: Seasonal Influenza vaccine
- Pregnant women: Pregnant women seasonal influenza vaccine
  Interventions: Biological: Seasonal Influenza vaccine
- Post partum women: Women who have given birth < 45 days seasonal influenza vaccine
  Interventions: Biological: Seasonal Influenza vaccine
- Children: Children from 6 months to 5 years of age seasonal influenza vaccine
  Interventions: Biological: Seasonal Influenza vaccine

INTERVENTIONS:
Biological: Seasonal Influenza vaccine — Seasonal Influenza vaccine
  Other Names: Flu vaccine

SUMMARY:
Rationale and background: Since 2013, IB has been performing passive pharmacovigilance activities related to TIV. Objetive: To implement an active surveillance study as part of our pharmacovigilance plan while passive surveillance activities will continue. Pharmacovigilance data on TIV, via active surveillance, is being implemented in response to WHO requirements for pre-qualification of TIV.

Study Design: This is a prospective cohort study. Population: Target groups for vaccination defined by The National Immunization Program of Brazil: children between six months and five years old; pregnant women; postpartum women (mothers until 45 days after birth); healthcare workers; and elderly (people over 60 years old). Study Size: A total of 900 individuals (300 health care workers, 300 elderly, 100 pregnant women, 100 post-partum women and 100 children between six months and five years old), presenting for immunization with IB TIV, and who agree to participate after providing Informed Consent.

Data Analyses: Descriptive approaches will be used to meet the defined objectives described in the protocol, as well as formal statistical tests when appropriate.

DETAILED DESCRIPTION:
Primary objective: to characterize and estimate the incidence of solicited adverse events following immunization (AEFI) associated with administration of the trivalent influenza vaccine produced at Butantan Institute (TIV).

Secondary objectives: 1) to characterize and estimate the incidence of overall (solicited and unsolicited) AEFI associated with administration of TIV; 2) to characterize and estimate the incidence of unsolicited AEFI associated with administration of TIV.

Study Design: This is a prospective cohort study aimed at identifying and evaluating adverse events following immunization among individuals vaccinated with TIV during the national immunization campaign. The design will include active surveillance by phone contact and through visits to the study site. Health facilities will be designated and set up as sentinel sites to enroll individuals being vaccinated with IB TIV for active follow up of solicited AEFI occurring within the first 14 days post-vaccination, and unsolicited AEFI up to 6 weeks post-vaccination.

Population: The following groups are targeted groups for the national immunization campaign and will be recruited for participation in this study:

* children between six months and five years old;
* pregnant women; postpartum women (mothers until 45 days after birth);
* healthcare workers; and
* elderly (people over 60 years old).

Variables: Solicited AEFI to be monitored will include local reactions (erythema, pain, swelling, ecchymosis, pruritus and induration), systemic reactions (headache, fever, malaise, arthralgia, myalgia, rash, chills, pruritus, fatigue, sweating) and irritability and persistent crying (for children than 6 years). Unsolicited AEFI reported over the period up to 6 weeks post-vaccination will be recorded. All adverse events reported in the study will be MedDRA coded. Other variables of interest in the study are demographic information of study participants: date of birth, gender, age, ethnicity, as well as vaccination information including date of immunization, site, and vaccine lot.

Data Sources: Study information including signs and symptoms following immunization with TIV will be recorded daily for 14 days post immunization, and will be recorded in the participant's study file.

Study Size: A total of 900 individuals (300 health care workers, 300 elderly, 100 pregnant women, 100 post-partum women and 100 children between six months and five years old), presenting for immunization with IB TIV, and who agree to participate after providing Informed Consent, will be enrolled in the study by study staff.

Data Analyses: Descriptive approaches will be used to meet the defined objectives described in the protocol, as well as formal statistical tests when appropriate. Incidence rates (IR) of AEFI with TIV will be calculated as the number of events divided by the total number of participants exposed to TIV in each of the targeted groups over the period of follow up. IR will be calculated based on total person time of follow-up, 95% confidence intervals will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Children between six months and five years old; or
* Pregnant and postpartum women (mothers until 45 days after birth); or
* Health care workers; or
* Elderly (aged 60 years or more); and
* To have indication to be vaccinated against influenza;
* To be available to participate in the study throughout its duration (6 weeks after any vaccine dose administered); and
* Demonstrates interest to participate in the study as registered in the informed consent form (ICF).

Exclusion Criteria:

* Known systemic hypersensitivity to eggs or to any component of the vaccine;
* Suspected or confirmed fever in the 3 days prior to vaccination or axillary temperature greater than 37.8 ° C on the day of vaccination;
* History of severe adverse reaction after previous administration of an Influenza vaccine within 6 weeks following vaccination;
* History of Guillain-Barre Syndrome or other demyelinating disease;
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
* Any other condition in the opinion of the investigator that justifies exclusion from participation.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: People eligible for immunization with seasonal influenza vaccine as described: children aged 6m-5y, elderly, health care workers, pregnant and post partum women.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute | study period follow up, approximately 6 months
  Solicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute

SECONDARY OUTCOMES:
Solicited and unsolicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute | study period follow up, approximately 6 months
  Solicited and unsolicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute
Unsolicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute | study period follow up, approximately 6 months
  Unsolicited adverse events following immunization with trivalent influenza vaccine produced by Butantan Institute

CONTACTS AND LOCATIONS:
Overall Officials: Lily Weckx, MD, Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - UBS Buritis, Boa Vista, Roraima
  - Crie - Unifesp, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gattas VL, Braga PE, Koike ME, Lucchesi MBB, Oliveira MMM, Piorelli RO, Queiroz V, Precioso AR. Safety assessment of seasonal trivalent influenza vaccine produced by Instituto Butantan from 2013 to 2017. Rev Inst Med Trop Sao Paulo. 2018 Dec 20;61:e4. doi: 10.1590/S1678-9946201961004. PMID 30570077